CLINICAL TRIAL: NCT06608030
Title: Effect of a Single Dose of Esketamine on Perioperative Negative Mood in Patients Undergoing Cardiac Valve Surgery: a Randomized Controlled Trial
Brief Title: Effect of Esketamine on Perioperative Negative Mood in Patients Undergoing Cardiac Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); The Sixth Medical Center of Chinese PLA General Hospital (Unknown)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLAGH-RCT-Esket
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Depression, Anxiety; Cardiac Surgery; S-ketamine
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): Patients who undergo general anesthesia using esketamine.
  Interventions: Drug: Esketamine
- Control group (Placebo Comparator): Patients who undergo general anesthesia without esketamine
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esketamine — A single dose of 0.3mg / kg esketamine during induction of anesthesia.
  Arms: Esketamine group
Drug: normal saline — Receiving the same volume of normal saline during induction of anesthesia.
  Arms: Control group

SUMMARY:
A multicenter, randomized controlled, blinded prospective study to investigate the effects of esketamine on perioperative anxiety and depression in patients undergoing cardiac valve surgery.

DETAILED DESCRIPTION:
Undergoing surgery can be a traumatic and painful experience for patients, often causing negative moods such as anxiety and depression. The size and type of surgery significantly impact the occurrence of anxiety and depression in patients. Approximately one-third of patients after cardiac surgery experience anxiety or depression, which increases the risk of recurrent cardiovascular events and death.

Ketamine is an anesthetic drug with comprehensive effects, including analgesia, sedation, and amnesia. Its primary mechanism of action is blocking N-methyl-D-aspartate (NMDA) receptors. Esketamine, the pure dextro isomer of ketamine, has a higher affinity for glutamate NMDA receptors and opioid receptors, offering stronger sedative, analgesic, and antidepressant effects. On March 4, 2019, esketamine was approved by the FDA for treatment-resistant depression. Given its analgesic, anesthetic, and antidepressant effects, esketamine may be an ideal drug for improving negative moods in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female
2. Patients undergoing heart valve surgery
3. Patients with ASA grade 1 to 4
4. BMI between 18-30 kg/m²
5. Able to participate in neuropsychological testing and receive follow-up visits
6. Clearly understand and voluntarily agree to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Patients with significant preoperative neuro-psychiatric disease and cognitive impairment
2. Intellectual disability or a MiniMental State Examination (MMSE) score <24, or a speech disorder that may compromise their ability to undergo preoperative assessments
3. History of psychoactive drug abuse

5. Preoperative combined severe hepatic insufficiency or renal insufficiency 6. Any contraindications to ketamine or esketamine, such as refractory hypertension or hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Perioperative anxiety and depreession | Preoperative day 1, postoperative day 7 and day 30
  The primary outcomes were depression and anxiety, which were assessed using the Hospital Anxiety and Depression Scale (HADS). Perioperative anxiety was measured using the Hospital Anxiety and Depression Scale-Anxiety (HADS-A) subscale, a standardized self-report instrument consisting of 7 items. Patients with a HADS-A score of 8 or more were considered to be experiencing anxiety, with a score of 8 to 10 indicating mild anxiety, 11 to 14 indicating moderate anxiety, and 15 to 21 indicating severe anxiety. Perioperative depression was measured using the Hospital Anxiety and Depression Scale-Depression (HADS-D) subscale. Patients with a HADS-D score of 8 or more were considered to be experiencing depression, with a score of 8 to 10 indicating mild depression, 11 to 14 indicating moderate depression, and 15 to 21 indicating severe depression.

SECONDARY OUTCOMES:
Postoperative Sleep Quality | Preoperative day 1, postoperative day 7 and day 30
  Postoperative sleep quality was assessed using the Insomnia Severity Index (ISI). The ISI is a simple tool used to screen for insomnia and consists of 7 items to assess the nature and symptoms of the subject's sleep disorder on a 5-point Likert scale, with each item scored from 0 to 4 and the total score ranging from 0 to 28, with higher scores indicating greater severity of insomnia. The sum of the scores with 0-7 indicating insomnia without clinical significance, 8-14 indicating subclinical insomnia, 15-21 indicating clinical insomnia (moderate), 22-28 indicating 'clinical insomnia (moderate), and 22-28 indicating clinical insomnia (moderate). A score of 8 to 14 indicates subclinical insomnia, a score of 15 to 21 indicates clinical insomnia (moderate), and a score of 22 to 28 indicates clinical insomnia (severe).
Delirium | Within 7 days after surgery
  Delirium was assessed using a combination of the 3-Minute Diagnostic Interview for CAM (3D-CAM) and the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Patients in the general ward were assessed using the 3D-CAM, while patients in the intensive care unit were assessed using the CAM-ICU. Delirium consists of four main features: acute altered mental status or fluctuating level of consciousness, inattention, disorganized thinking, and altered level of consciousness. Patients were diagnosed with postoperative delirium if both the first and second features were present, and either the third or fourth feature was also present.
PONV | Within 2 days after extubation
  Postoperative nausea and vomiting (PONV) were assessed using a visual analogue scale (VAS). This scale consists of a 10-centimeter straight line, with 0 indicating no nausea and vomiting, and 10 indicating the most extreme level of nausea and vomiting that can be endured. The severity of PONV is categorized as follows: mild (1 to 4), moderate (5 to 6), and severe (7 to 10).
Postoperative Recovery Quality | Postoperative day 7 and day 30
  Postoperative quality of recovery was evaluated using the Chinese version of the Quality of Recovery-15 (QoR-15) score. This assessment tool comprises 15 items, each scored on a 10-point scale. The total score ranges from 0 to 150, with 0 indicating poor recovery and 150 signifying an excellent quality of recovery.
Postoperative Pain | Postoperative day 7 and day 30
  Assessment was conducted using the Numerical Rating Scale (NRS) for pain, which ranges from 0 to 10. On this scale, a score of 0 represents the absence of pain, while a score of 10 represents the most severe pain.
Postoperative Quality of Life | Postoperative day 7 and day 30
  Postoperative quality of life was evaluated using the EQ-5D, a five-dimensional health scale. This scale encompasses five key dimensions: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension is rated on a three-point scale: no difficulty, some difficulty, and extreme difficulty. The responses to these levels are then utilized to calculate the EQ-5D Index score, which quantifies the overall health status based on the reported levels of difficulty across the five dimensions.

OTHER OUTCOMES:
Intraoperative blood pressure | During the surgery
  Intraoperative blood pressure（MAP in mmHg/SBP in mmHg/DBP in mmHg) at T0 (before induction of anes thesia), T1 (5 min after esketamine or control injection), T2 (30 min after esketamine or control injection), T3 (1 h after esketamine or control injection), T4 (3 h after esketamine or control injection), and T5(at the end of surgery) were included.
Intraoperatively heart rate | During the surgery
  Intraoperative heart rate（HR in bmp) at T0 (before induction of anes thesia), T1 (5 min after esketamine or control injection), T2 (30 min after esketamine or control injection), T3 (1 h after esketamine or control injection), T4 (3 h after esketamine or control injection), and T5(at the end of surgery) were included.
Perioperative inflammatory factor (IL-6) | perioperatively
  Inflammatory factor (IL-6 in pg/ml) were from laboratory tests in the patient's medical record.
Perioperative inflammatory factor (CRP) | perioperatively
  Inflammatory factor (CRP in mg/dl) were from laboratory tests in the patient's medical record.
Perioperative brain injury-related factor (S100β) | perioperatively
  Brain injury-related factor (S100β in ng/ml)
Perioperative brain-derived neurotrophic factor (BDNF) | perioperatively
  Brain-derived neurotrophic factor (BDNF in ng/ml)
Perioperative acetylcholine (Ach) | perioperatively
  Acetylcholine (Ach in ng/ml)
Perioperative norepinephrine (NE) | perioperatively
  Norepinephrine(NE in ng/ml)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Medical center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang ZN, Hao XY, Cai C, Sun L, Zhang ZY, Wang M, Wu YS, Wang Y, Cao JB, Liu YH, Lou JS, Fu Q, Jiang SL, Han RQ, Mi WD, Tong L. Effect of esketamine on postoperative depression and anxiety in patients undergoing cardiac valve surgery: A randomised, placebo-controlled, double-blinded clinical trial. Pharmacol Res. 2025 Dec;222:108047. doi: 10.1016/j.phrs.2025.108047. Epub 2025 Nov 22. PMID 41285329